CLINICAL TRIAL: NCT05021796
Title: Telecounselling as a Virtual Platform to Replace On-the-job Training for Asthma Counseling
Brief Title: Telecounselling for Asthma Counseling
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Mei Fong Liew, Consultant, Division of Respiratory & Critical Care Medicine, National University Health System, Singapore
Other Study IDs: 2020/01460
Record Dates: First submitted 2021-08-15; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurses: Including criteria: (1) registered nurses, (2) nurses undergoing a training for asthma telecounseling, (3) age 21 or more.
  Excluding criteria: (1) nurses with previous training for asthma counseling, (2) nurses who do not take care of patients with asthma, (3) Pregnant women

SUMMARY:
In the coronavirus 2019 pandemic, on-the-job training for asthma counseling becomes more difficult. Telecounseling as a training platform becomes a mainstream of training during the pandemic. This study is designed to fill the knowledge gap for telecounseling as a training platform for asthma counseling among nurses.

DETAILED DESCRIPTION:
Asthma education is essential in improving outcomes in asthma management. Patients with asthma exacerbation frequently present to the urgent care centre or emergency department for emergency treatment. Nurse-led asthma education was considered as beneficial to asthma management. However, not all nursing staff in the urgent care centre and emergency department are equipped with skills to counsel patients regarding their asthma control and inhaler use. It is important to empower the nursing staff with these skills such that the care of patients with asthma is not compromised.

In the coronavirus 2019 pandemic, on-the-job training for asthma counseling becomes more difficult. Asthma counseling trainers were usually in the clean zones but recipients of asthma counseling training were usually in the dirty zones. Telecounseling as a training platform becomes a mainstream of training during the pandemic. Telehealthcare interventions on patients with asthma was proven to reduce hospitalization over a 12-month period in a previous meta-analysis. However, there was no study investigating the efficacy of telecounseling to replace on-the-job training for asthma counseling. This study is designed to fill the knowledge gap for telecounseling as a training platform for asthma counseling among nurses.

ELIGIBILITY:
Including criteria:

* registered nurses
* nurses undergoing a training for asthma telecounseling
* age 21 or more.

Excluding criteria:

* nurses with previous training for asthma counseling
* nurses who do not take care of patients with asthma
* Pregnant women

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is to investigate the efficacy of telecounseling to replace on-the-job training for asthma counseling. This study is designed to fill the knowledge gap for telecounseling as a training platform for asthma counseling among nurses. Hence, the study population consists of nurses who are new to asthma counseling.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy on asthma teaching scale | Immediately before and immediately after the telecounseling training
  Chiang LC, Hsu JY, Liang WM, Yeh KW, Huang JL. Developing a scale to measure self-efficacy on asthma teaching for health care providers. J Asthma. 2009;46(2):113-117.

SECONDARY OUTCOMES:
Satisfaction of the training | Immediately after the telecounseling training
  Satisfaction of the training
Qualitative data - Focused Interview with the following specific open-ended questions | Immediately after the telecounseling training
  1. What did participants learn from attending Telecounselling?
  2. Are participants more confident in carrying out asthma counselling after attending telecounselling? And why?
  3. Will participants recommend this mode of learning/modelling be added on to future education initiatives on counselling?
  4. Any other good points about this experience?
  5. Any bad points about this experience?

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali A, Pena SG, Huggins C, Lugo F, Khaja M, Diaz-Fuentes G. Impact of Group Asthma Education on Asthma Control and Emergency Room Visits in an Underserved New York Community. Can Respir J. 2019 Oct 1;2019:5165189. doi: 10.1155/2019/5165189. eCollection 2019. PMID 31662806
- [Background] Frey SM, Contento NC, Halterman JS. Nurse-delivered outpatient asthma education for children and caregivers: a pilot study to promote shared asthma management. J Asthma. 2021 Mar;58(3):413-421. doi: 10.1080/02770903.2019.1692028. Epub 2019 Nov 18. PMID 31739709
- [Background] Spaggiari S, Gehri M, Di Benedetto L, Hafen GM, Pauchard JY, Gervaix A, Pannatier A, Sadeghipour F, Di Paolo ER. Inhalation technique practical skills and knowledge among physicians and nurses in two pediatric emergency settings. J Asthma. 2021 Feb;58(2):190-196. doi: 10.1080/02770903.2019.1674329. Epub 2019 Oct 17. PMID 31566459
- [Background] McLean S, Chandler D, Nurmatov U, Liu J, Pagliari C, Car J, Sheikh A. Telehealthcare for asthma. Cochrane Database Syst Rev. 2010 Oct 6;2010(10):CD007717. doi: 10.1002/14651858.CD007717.pub2. PMID 20927763
- [Background] Chiang LC, Hsu JY, Liang WM, Yeh KW, Huang JL. Developing a scale to measure self-efficacy on asthma teaching for health care providers. J Asthma. 2009 Mar;46(2):113-7. doi: 10.1080/02770900802444245. PMID 19253113